CLINICAL TRIAL: NCT00822627
Title: Influenza Vaccination in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Katherine M Hiller, MD, Department of Emergency Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Influenza
Keywords: Influenza; vaccination; Emergency Department
MeSH Terms: conditions — Influenza, Human; Emergencies | interventions — Influenza Vaccines; Educational Status; Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccination group (Experimental): Vaccination group
  Interventions: Drug: Influenza Vaccination
- Education/referral (Experimental): Education/referral
  Interventions: Behavioral: Education and referral

INTERVENTIONS:
Drug: Influenza Vaccination — 0.5 mL Sanofi-Pasteur intramuscular influenza vaccination
  Arms: Vaccination group
Behavioral: Education and referral — Patients are given information regarding the inactivated influenza vaccination and a list of community providers who provide influenza vaccination
  Arms: Education/referral

SUMMARY:
Randomized controlled trial of influenza vaccination versus referral for vaccination in the Emergency department. Is the Emergency Department an effective venue for vaccination for influenza? Does vaccination for influenza in the Emergency Department change the rates of influenza, influenza-like-illness or medical provider visits when compared with patient referred for vaccination in the community?

DETAILED DESCRIPTION:
This study is a prospective randomized, controlled trial of influenza vaccination vs referral for influenza vaccination in the Emergency Department. Subjects are either offered vaccination or education regarding vaccination and a list of community providers. At a four-month follow up, rates of influenza, influenza-like illness and number of medical provider visits are determined.

ELIGIBILITY:
Inclusion Criteria:

* Unvaccinated patients presenting to the Emergency Department aged 6 months or more who have at least one high risk attribute:
* Age 6-59 months or >50 years
* Pregnant
* Health care worker
* Aged 6 months-18 years on chronic aspirin therapy
* Comorbidity (cardiovascular disease, pulmonary disease, metabolic disease, renal disease, hepatic disease, seizures, neuromuscular disease, cognitive dysfunction, or any reason to have had regular medical follow up or hospitalization in the preceding year)
* Household contact or caregiver of someone with at least one high risk attribute

Exclusion Criteria:

* Prior vaccination
* History of Guillan-Barre syndrome within 6 weeks of prior influenza vaccination
* Allergy to influenza vaccination or eggs
* Age < 6 months old
* Fever with more than minor illness
* Hospitalization

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Vaccination status | 4 months

SECONDARY OUTCOMES:
Influenza rate | 4 months
Influenza-like illness rate | 4 months
Visits to medical providers | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Hiller, MD, Principal Investigator — University of Arizona Department of Emergency Medicine
Locations (1):
- University of Arizona, Tucson, Arizona, United States